CLINICAL TRIAL: NCT03373097
Title: Phase I/II Study of Anti-GD2 Chimeric Antigen Receptor-Expressing T Cells in Pediatric Patients Affected by High Risk and/or Relapsed/Refractory Neuroblastoma or Other GD2-positive Solid Tumors
Brief Title: Anti-GD2 CAR T Cells in Pediatric Patients Affected by High Risk and/or Relapsed/Refractory Neuroblastoma or Other GD2-positive Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Franco Locatelli, Haematology-Oncology Department Chief, Bambino Gesù Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD2CAR01
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma; Neuroblastoma Recurrent; GD2-positive Solid Tumors; Osteosarcoma; Ewing Sarcoma; Sarcoma
Keywords: Neuroblastoma; GD2 CAR T cell; CAR T; GD2-positive solid tumors; Osteosarcoma; Ewing Sarcoma; GD2-positive sarcoma
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma; Sarcoma, Ewing; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GD2-CART01 (Experimental): After a lymphodepleting regimen the patients will receive 1.0 to 10.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells.
  Interventions: Biological: GD2-CART01

INTERVENTIONS:
Biological: GD2-CART01 — Following a lymphodepleting treatment with conventional chemotherapy, patients will be treated with 1.0 to 10.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.

SUMMARY:
The purpose of this study is to test the safety and efficacy of GD2-CART01, a CAR T cell treatment targeting GD2 in paediatric or young adult patients with High Risk and/or relapsed/refractory Neuroblastoma.

A small exploratory cohort of patients with GD2-positive tumors other than Neuroblastoma has also been included.

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I or dose escalation phase and a Phase II or expansion phase. Paediatric or young adult patients with relapsed High Risk and/or relapsed/refractory Neuroblastoma will be enrolled in the study.

After completion of the phase I portion of the study, a small cohort of patients with GD2-positive tumors other than Neuroblastoma has also been included.

Eligible patients will undergo leukapheresis in order to harvest T cells, which will be manufactured to obtain the autologous CAR T product GD2-CART01, a GD2-targeting CAR T product. Briefly, the patients will be treated with a lymphodepleting regimen containing conventional chemotherapic agents and subsequently will receive a single infusion of GD2-CART01. Moreover, the product contains a suicide gene safety switch (namely inducible Caspase 9): in case of relevant toxicities, the patient will receive the dimerizing agent in order to activate the apoptotic pathway in the infused T cells.

After infusion of CAR T cells, the patients will enter a 5-year active follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Phase I The patient must meet the following eligibility inclusion criteria to be enrolled to receive treatment in the Phase I study.

1. Diagnosis of NBL that have been treated with frontline therapy and is judged to be incurable, based upon the following criteria:

   1. Relapse after first-line treatment, proved by a positive 123-I-mMIBG-scan
   2. Persistence/progression of disease after the initiation of the upfront treatment
2. Patients must have measurable or evaluable disease at the time of treatment enrollment, as shown by bone marrow biopsy/aspirate, US or CT/MRI scan or by 123-I-mMIBG scan.
3. Recover from the toxic effect of previous chemotherapies: grade 4 and or 3 non-hematologic toxicities must have resolved to grade ≤2; if some effects of the therapies have become chronic (i.e. treatment associated thrombocytopenia), the patient must be clinically stable, according to the opinion of the treating physicians, and meet all other eligibility criteria.
4. Age: 12 months -18 years.
5. Voluntary informed consent is given. For subjects < 18 years old their legal guardian must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
6. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients less than or equal to 16 years of age: Lansky scale greater than or equal to 60%.
7. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
8. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.

Phase II

The patient must meet the following eligibility inclusion criteria to be enrolled to receive treatment in the Phase II study.

1. Diagnosis of NBL that have been treated with frontline therapy and is judged to be incurable, based upon the following criteria:

   1. Relapse after first-line treatment, proved by a positive MIBG-scan
   2. Persistence/progression of disease after the initiation of the upfront treatment

   OR
2. Diagnosis of extremely High Risk NBL at high risk of relapse, defined by stage III/IV and Myc-N amplification, at the end of the first-line treatment according to the Standard of Care, even if NED.

   OR
3. Diagnosis of GD2+ tumors other than Neuroblastoma, considered incurable with conventional treatments by the treating physician.
4. Patients with relapsed/refractory disease must have measurable or evaluable disease at the time of treatment enrollment, as shown by bone marrow biopsy/aspirate, US or CT/MRI scan or by MIBG-scan.
5. Recover from the toxic effect of previous chemotherapies: grade 4 and or 3 non-hematologic toxicities must have resolved to grade ≤2; if some effects of the therapies have become chronic (i.e. treatment associated thrombocytopenia), the patient must be clinically stable, according to the opinion of the treating physicians, and meet all other eligibility criteria.
6. Age: 12 months - 18 years.
7. Voluntary informed consent is given. For subjects < 18 years old their legal guardian must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
8. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients less than or equal to 16 years of age: Lansky scale greater than or equal to 60%.
9. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
10. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe, uncontrolled active intercurrent infections
3. Active hepatitis B or hepatitis C infection
4. HIV infection
5. Rapidly progressive disease with life-expectancy < 6 weeks
6. History of grade 3 or 4 hypersensitivity to murine protein-containing products
7. Hepatic function: Inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6 x ULN based on age and laboratory specific normal ranges
8. Renal function: serum creatinine > 3x ULN for age.
9. Blood oxygen saturation < 90%.
10. Cardiac function: Left ventricular ejection fraction lower than 45% by ECHO.
11. Marrow function: ANC lower than 500/mm3 and/or platelets lower than 20.000 (not reached by transfusion).
12. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject.
13. Untreated CNS metastasis; patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
14. Concurrent or recent prior therapies, before infusion:

    1. Systemic steroids (at a dose equivalent to or greater 2 mg/kg prednisone) in the 2 weeks before infusion. Recent or current use of inhaled/topical/non-absorbable steroids is not exclusionary.
    2. Systemic chemotherapy in the 2 weeks preceding infusion.
    3. Immunosuppressive agents less than or equal to 30 days.
    4. Radiation therapy must have been completed at least 3 weeks prior to enrollment.
    5. I131-MIBG therapy must have been completes at least 6 weeks prior to enrollment
    6. Anti-GD2 murine monoclonal antibody (ch14.18 antibody) in the 2 weeks preceding infusion
    7. Other anti-neoplastic investigational agents currently or within 30 days prior to start of protocol therapy;
    8. Exceptions:
    9. Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis
15. Patient-derived GD2-CART01 production failure.

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase I - Identification of the dose limiting toxicity (DLT) | 4 weeks after T cell infusion
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 4 and the number of patients experiencing DLT will be evaluated
Phase II - Antitumor effect | Up to 6 months after T cell infusion
  Assessment of Best Overall Response (BOR)

SECONDARY OUTCOMES:
In vivo persistence/expansion of infused CAR T cell | UP to 5 years
  Detection of infused CAR T cell in the peripheral and bone marrow blood
Serum cytokine profiling | First 2 weeks after T cell infusion
  Assessment of the seric cytokines profile
Time To Progression (TTP) | Up 5 years after T cell infusion
Event-Free Survival (EFS) | Up 5 years after T cell infusion
Overall Survival (OS) | Up 5 years after T cell infusion
Disease outcome according to INRC vs irRC | Up to 5 years
  Tumor response assessment through the two different criteria
Elimination of CAR T cell through iC9 in case of toxicity | Up to 15 years
  Assessment of the kinetic of CAR T cell elimination after infusion of the dimerizer

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Locatelli F, Pagliara D, De Ioris MA, Becilli M, Del Baldo G, Serra A, Mastronuzzi A, Cefalo MG, Li Pira G, Leone G, Bertaina V, Fabozzi F, Di Nardo M, Rosignoli C, D'Andrea ML, Crocoli A, Vennarini S, Sinibaldi M, Di Cecca S, Guercio M, Iaffaldano L, Lucarelli B, Algeri M, Merli P, Colafati GS, De Angelis B, Quintarelli C, Del Bufalo F. GD2-targeting CAR T cells in high-risk neuroblastoma: a phase 1/2 trial. Nat Med. 2025 Nov;31(11):3689-3699. doi: 10.1038/s41591-025-03874-6. Epub 2025 Aug 21. PMID 40841488
- [Derived] Yeku OO, Longo DL. CAR T Cells for Neuroblastoma. N Engl J Med. 2023 Apr 6;388(14):1328-1331. doi: 10.1056/NEJMe2300317. No abstract available. PMID 37018497
- [Derived] Del Bufalo F, De Angelis B, Caruana I, Del Baldo G, De Ioris MA, Serra A, Mastronuzzi A, Cefalo MG, Pagliara D, Amicucci M, Li Pira G, Leone G, Bertaina V, Sinibaldi M, Di Cecca S, Guercio M, Abbaszadeh Z, Iaffaldano L, Gunetti M, Iacovelli S, Bugianesi R, Macchia S, Algeri M, Merli P, Galaverna F, Abbas R, Garganese MC, Villani MF, Colafati GS, Bonetti F, Rabusin M, Perruccio K, Folsi V, Quintarelli C, Locatelli F; Precision Medicine Team-IRCCS Ospedale Pediatrico Bambino Gesu. GD2-CART01 for Relapsed or Refractory High-Risk Neuroblastoma. N Engl J Med. 2023 Apr 6;388(14):1284-1295. doi: 10.1056/NEJMoa2210859. PMID 37018492
- [Derived] Tumino N, Weber G, Besi F, Del Bufalo F, Bertaina V, Paci P, Quatrini L, Antonucci L, Sinibaldi M, Quintarelli C, Maggi E, De Angelis B, Locatelli F, Moretta L, Vacca P, Caruana I. Polymorphonuclear myeloid-derived suppressor cells impair the anti-tumor efficacy of GD2.CAR T-cells in patients with neuroblastoma. J Hematol Oncol. 2021 Nov 12;14(1):191. doi: 10.1186/s13045-021-01193-0. PMID 34772439